CLINICAL TRIAL: NCT06681545
Title: An Exploration of the Experiences and Support Needs of Young Adults With Severe and Uncontrolled Asthma
Brief Title: Exploring the Lived Experience of Young Adults With Severe Asthma
Acronym: EaSY
Status: Recruiting | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: Burdett Trust for Nursing (Other); Liverpool University Hospitals NHS Foundation Trust (Other Government); University of Manchester (Other)
Responsible Party: Sponsor
Other Study IDs: B02178
Record Dates: First submitted 2024-10-22; First posted 2024-11-08 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Asthma; Severe Asthma; Uncontrolled Asthma
Keywords: young people; young adults; young person
MeSH Terms: conditions — Asthma | interventions — Focus Groups

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- young adults with severe and or uncontrolled asthma: no intervention to be administered. Participants will be asked to participate in 1-1 interviews and or focus group interviews
  Interventions: Other: one to one interviews and or focus groups

INTERVENTIONS:
Other: one to one interviews and or focus groups — one to one interviews and or focus groups

SUMMARY:
Asthma is a serious long-term lung condition caused by swollen airways that narrow. This causes wheezing, chest tightness, and breathlessness. Most asthma is well-controlled with medication.

However, 5-10% of asthmatics have severe asthma where treatment does not control symptoms and up to 67% of asthmatics have uncontrolled asthma, caused by not always taking medication as recommended, lifestyle choices or other health problems worsening their asthma.

In the UK, asthma affects around 800,000 young adults. This group is at high-risk of having poor asthma control, worse outcomes than other age-groups. This is because young adults need care that differs from other age-groups and current care is not meeting these needs.

There is little information on the experiences and needs of this group and very few studies exist, exploring how to improve care. This study will explore the experiences and needs of young adults (age16-25) with severe and uncontrolled asthma.

Methods. The investigators will perform two study-arms with young adults with severe/uncontrolled asthma in Manchester and Liverpool severe asthma centres:

Study-arm 1: Interview participants using photographs chosen by them to help explain their experiences of living with asthma and support that they need.

Study arm 2: Perform group interviews to understand participants' thoughts around the insights from study-arm 1 combined with their own experiences. To explore and develop ideas on how to improve future care.

At the end of both study arms, a workshop involving patients and stakeholders involved in delivering care will take place, to identify a joint goal of how to improve care in this cohort and map ways in which to achieve this.

Together, the study results and workshop will increase our understanding of the experiences and needs of young adults with asthma. Helping us to identify new ways to improve care which can be tested in future research.

DETAILED DESCRIPTION:
Research question "What are the experiences, and support needs of young adults living with severe and uncontrolled asthma?"

Aim To develop a rich in-depth understanding of the lived experiences, challenges, and perceived support needs of being a young adult with severe and or uncontrolled asthma.

Objectives

1. Examine in -depth the day-to-day experiences of living with severe asthma through undertaking 1-1 in-depth interviews using photo elicitation techniques.
2. Identify participant support needs through undertaking focus groups
3. Combine results from 1-1 and focus group interviews, to help inform and develop future interventions/research.
4. To develop a theory of change with patients and stakeholders.

Study design A qualitative design using photo elicitation driven semi-structured one-to-one interviews (work package 1) followed by focus group interviews, (work package 2) concluding with a Theory of Change (TOC) workshop.

Data collection Work package 1: In-depth interviews - Post consent participants will be asked to select/take and bring between 3-5 pictures or self-taken photographs to the 1-1 interview to help them describe their experiences of living with asthma to the interview. The interviews will be conducted using a pre-designed semi-structured interview schedule and the participant's selected images to guide the interview. Interviews can be either face-to-face in person or online via MS subject to participant choice. The interviews will be audio recorded and uploaded post interview.

Demographic details (age, gender, ethnicity, and educational attainment) and medical history will be obtained from within the medical records, by the PI including Asthma Phenotype, Medication use, Lung function/FeNO and recent ACQ/AQLQ questionnaire results and completed onto a Case report form.

Work package 2: Focus groups - There will be two separate focus groups of between 4-8 participants. They will be face-to-face with the focus groups being led by the PI and supported by a PPIE engagement officer. The focus groups will be audio recorded on an encrypted dictaphone for future transcription. The focus groups will start with a summary of the results derived from the1-1 interviews and a synopsis of previous interventions to date in other research. the investigators will ask participants to consider their own support needs and to provide suggestions for future care interventions within the focus groups. Participant medical history and demographic details (age gender, ethnicity and educational attainment) will be obtained from within the medical notes by the PI.

A TOC workshop will assemble patients and stakeholders involved in the receipt and delivery of care of young adults with severe and uncontrolled asthma and will be facilitated to develop a 'theory-of-change'. The output of the TOC meeting will be a TOC process map and a detailed report of all discussions.

Statistical analysis Demographic and clinical data will be presented descriptively using appropriate statistics, including mean (standard deviation), median (interquartile range), N (percentage), and graphics.

Qualitative data analysis The in-depth 1-1 interviews will be analysed using interpretive phenomenological analysis, whereas the focus groups will be analysed using thematic analysis.

Research Ethics Committee (REC) Before the start of the study, a favourable opinion will be sought from a REC and HRA for the study protocol, informed consent forms and other relevant patient facing documents.

Patient & Public Involvement This proposed research has been amended and refined over the last four years with young adults. Within this research the investigators will work with a Patient and Public engagement officer and Patient Advisory Group (PAG) consisting of 3-5 individuals to advise on many elements of the study.

Dissemination On completion of the study a final study report will be prepared. It is also intended to publish the results from both work packages in peer reviewed journal's, be presented at professional conference and submitted as part of a PhD thesis.

A study summary leaflet will be designed for both work packages The thematic content of the in-depth interviews and participant photographs/pictures (Subject to opting in on the consent form) will be developed into a short creative media video, outlining the results in a manner understandable for the lay public. The in-depth interviews and focus groups combined will also be made into a short media illustration to facilitate easy understanding by the lay public.

ELIGIBILITY:
Inclusion Criteria:

* A confirmed diagnosis of severe or uncontrolled asthma under the care of the Manchester or Liverpool severe asthma services
* Participants aged 16-25 years.
* Informed consent provided.

Exclusion Criteria:

* Inability to provide informed consent.
* Participants with additional long-term conditions who identify their dominant health concern to be non-asthma related.
* Focus group only- inability to converse in English

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: young adults age 16-25 with severe or uncontrolled asthma
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Patient perceived experiences and challenges of living with severe and or uncontrolled asthma | 12 months
  The investigators are not directly using tools/scales to measure outcome measures but will be using the data generated from the in depth interviews and focus groups to understand subjective participant perceived experiences and challenges of living with severe/uncontrolled asthma. in seeking to understand this, the investigators will meet the intended primary outcomes of the study.

OTHER OUTCOMES:
patient perceived support needs | 12 months
  The investigators will not be using scales or tools to measure outcomes, but will be using the in-depth interviews and focus groups to understand participants subjective perceived support needs, in seeking to understand this, the investigators will meet the intended outcomes of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Severe asthma services based at both Manchester University Foundation NHS trust and Liverpool University Foundation NHS Trust, Manchester, Greater, United Kingdom

IPD SHARING:
Plan to Share IPD: No